CLINICAL TRIAL: NCT00147875
Title: PVAG - Phase I/II Dose Finding Trial in Elderly Patients (> 60 Years) With Advanced Stages Hodgkin's Lymphoma
Brief Title: Study of Prednisone, Vinblastine, Doxorubicin, and Gemcitabine in Elderly Patients With Advanced Stages Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: German Hodgkin's Lymphoma Study Group (Other); Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PVAG elderly
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2009-09-07 (Estimated); Status verified 2009-09

CONDITIONS: Hodgkin's Disease
Keywords: Lymphoma; Gemcitabine; Advanced stages Hodgkin's lymphoma; Elderly
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Prednisone; Vinblastine; Doxorubicin; Gemcitabine

INTERVENTIONS:
Drug: Prednisone
Drug: Vinblastine
Drug: Doxorubicin (Adriamycin)
Drug: Gemcitabine

SUMMARY:
The objectives of this study are to assess the feasibility and efficacy of a combination chemotherapy (PVAG) in elderly patients with advanced stages Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Gemcitabine shows promising activity in patients with relapsed lymphoma either administered as single agent or in combination with other cytotoxic agents. No trial to date evaluated its role in patients with primary Hodgkin's lymphoma. We therefore developed a three-weekly regimen based on the standard ABVD regimen.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin's lymphoma (histologically proven)
* Clinical stage IIB (with risk factors bulky mediastinal mass and/or extranodal involvement), III, or IV
* No prior antitumor therapy
* Age 60 to 75 years
* WHO performance status 0-2
* Normal pulmonary function
* Written informed consent

Exclusion Criteria:

* The following histologies are excluded: lymphocyte predominant HD
* Leukocytes < 2,500/microL
* Platelets < 100,000/microL

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-03; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose-limiting toxicities and dose reductions
Phase II: Treatment administration and complete response rate

SECONDARY OUTCOMES:
Toxicities
Supportive care (RBCT need, antibiotic need)
Early progression rate
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Principal Investigator — University of Cologne
Locations (1):
- University of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Boll B, Bredenfeld H, Gorgen H, Halbsguth T, Eich HT, Soekler M, Markova J, Keller U, Graeven U, Kremers S, Geissler M, Trenn G, Fuchs M, von Tresckow B, Eichenauer DA, Borchmann P, Engert A. Phase 2 study of PVAG (prednisone, vinblastine, doxorubicin, gemcitabine) in elderly patients with early unfavorable or advanced stage Hodgkin lymphoma. Blood. 2011 Dec 8;118(24):6292-8. doi: 10.1182/blood-2011-07-368167. Epub 2011 Sep 13. PMID 21917759